CLINICAL TRIAL: NCT00397397
Title: Comparative Study in Patients With Lower Ureteral Stones Treated With 10 MG Alfuzosin,10 MG Alfuzosin With Rowatinex, and Rowatinex Alone
Brief Title: Comparative Treatment Study in Patients With Lower Ureteral Stones
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: 15/2006CTIL
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2006-11-09 (Estimated); Status verified 2006-11

CONDITIONS: Urinary Calculi
Keywords: Urinary Calculi; Rowatinex; Alfuzosin; Drug Therapy
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
We wish to determine the best treatment for expulsion of lower ureteral stones. Which of the three major treatment protocols is the best treatment of conservative management of ureteral stones?

DETAILED DESCRIPTION:
The study will include 60 patients with lower ureteral stones. The patients will be divided into three groups. The first group will be administered Alfuzosin (10 mg). The second group will be administered a combination of Alfuzosin (10 mg)and Rowatinex (Pinene 31%, Camphene 15%, Anetol 4%, Borneol 10%, Cineol 3%, Fenchenol 4%, Olive Oil 33%). The third group will be administered Rowatinex.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lower ureter (urinary calculi) up to 8mm
* Must be able to swallow tablets

Exclusion Criteria:

* Sensitivity to Alfuzosin and Rowatinex
* Pregnant and breastfeeding women
* Single kidney
* Obstructing stone
* Renal failure creatinine up to 1.8 mg/dl
* Patients using various alpha blockers
* Liver failure
* Fever higher than 38 C
* UTI
* Syncope or hypotension
* Patients treated with PDE5
* Patients treated with inhibitor CYP3A4
* Patients refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-01; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Faragi, Principal Investigator — Urology Department, Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel